CLINICAL TRIAL: NCT05853887
Title: iNUDGE: INtegration of liqUiD Biopsy Based Next Generation Gene sEquencing in Newly Diagnosed NSCLC - A Stepped Wedge Cluster Randomized Clinical Trial
Brief Title: Liquid Biopsy Based NGS in Newly Diagnosed NSCLC
Acronym: iNUDGE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Charu Aggarwal (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor-Investigator, Charu Aggarwal, Leslye M. Heisler Associate Professor of Lung Cancer Excellence and Associate Director, Penn Center for Precision Medicine, Abramson Cancer Center at Penn Medicine
Organization: Abramson Cancer Center at Penn Medicine (Other)
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: UPCC 27522; 852795 (Other: University of Pennsylvania Institutional Review Board)
Record Dates: First submitted 2023-04-07; First posted 2023-05-11 (Actual); Last update posted 2025-11-05 (Actual); Status verified 2025-11

CONDITIONS: Non Small Cell Lung Cancer Metastatic; Newly Diagnosed NSCLC; Non-Squamous Non-Small Cell Neoplasm of Lung
Keywords: Next Generation Sequencing; Liquid biopsy; Newly diagnosed; Molecular testing; Plasma based next generation sequencing; Electronic health record; Nudge intervention; Targeted therapy; Behavioral economics

STUDY DESIGN:
Intervention Model Description: This study employs a stepped-wedge cluster randomized clinical trial design. Randomization will occur at the group (site) level. Sites will be turned on according to the stepped-wedge cluster randomized design but will run in parallel.
Masking Description: This intervention is directed towards physicians. Individuals will not be randomized.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Penn Medicine New Jersey (Other): All sites with be randomized to implement the nudge at different points in time. Prospective data with be compared with each site's respective baseline numbers over a two-year period.
  Interventions: Behavioral: iNUDGE
- Penn Medicine Lancaster General Health (Other): All sites with be randomized to implement the nudge at different points in time. Prospective data with be compared with each site's respective baseline numbers over a two-year period.
  Interventions: Behavioral: iNUDGE
- Penn Presbyterian Medical Center (Other): All sites with be randomized to implement the nudge at different points in time. Prospective data with be compared with each site's respective baseline numbers over a two-year period.
  Interventions: Behavioral: iNUDGE

INTERVENTIONS:
Behavioral: iNUDGE — Electronic health record nudge which prompts physicians to order plasma-based NGS testing for eligible patients with newly diagnosed lung cancer.

SUMMARY:
This study expands the application of an electronic health record (EHR) "nudge" used to prompt physicians' clinical practice to order molecular testing at the time of initial diagnosis for patients with specific types of advanced lung cancer. The primary goal is to have these test results available prior to starting treatment so that physicians can make molecularly-informed treatment decisions. The second goal is to better understand factors that contribute to whether or not the EHR-nudge implementation is successful.

DETAILED DESCRIPTION:
At the University of Pennsylvania Health System (UPHS), a behavioral economics (BE) informed "nudge" strategy was piloted to guide physicians' clinical practice to include concurrent use of plasma and tissue-based next generation sequencing (NGS) testing at the time of initial diagnosis for patients with newly diagnosed metastatic non-squamous (mNSq) non-small cell lung cancer (NSCLC). These findings have demonstrated that behavioral, electronic health record (EHR)-based nudges are feasible and can promote guideline concordant diagnostic testing at both community and academic sites.

The overarching goal of this current trial is to expand the application of the BE informed nudges, which includes a Best Practice Advisory (BPA) and Electronic Decision Support Tool (e-CDS) approach, which has been operationalized within Epic, the EHR used at UPHS, to six satellite hospitals. Our central hypothesis is that this approach will dramatically increase adoption of comprehensive molecular testing and enhance the delivery of molecularly informed 1L therapy in patients with newly diagnosed mNSq NSCLC.

Intervention: A multicomponent BE-informed EHR-based nudge designed to facilitate comprehensive molecular testing by embedding a default P-NGS order into the EHR at the time of the NPV. If ordered, test results are incorporated into provider workflows and conveyed through electronic clinical decision support (e-CDS) notifications. This support program will notify clinicians of targetable mutations, potential clinical trials, as well as absence of mutations detected on plasma testing as a means of improving the timely delivery of molecularly informed therapy.

Study Design

Objective 1: In a stepped wedge cluster randomized trial of newly diagnosed patients with mNSq NSCLC, evaluate the effectiveness of a multicomponent BE-informed EHR-based nudge intervention at increasing timely receipt of comprehensive molecular test results prior to 1L therapy by incorporating P-NGS into the standard clinical workup.

The design of this trial will include 3 clusters, representing 6 community hospitals. There will be an initial period in which no clusters are exposed to the intervention. Subsequently, at regular intervals (the "steps") one cluster (or a group of clusters) will be randomized to cross from the control to the intervention under evaluation. This process will continue until all clusters have crossed over to be exposed to the intervention. At the end of the study there will be a period when all clusters are exposed. Data collection will continue throughout the study, so that each cluster will contribute observations under both control and intervention observation periods. Two years of baseline data will be obtained from all study sites for comparison.

Objective 2: Assess the contextual mechanisms influencing the adoption, reach, and effectiveness of EHR-based nudge interventions, with a lens for health equity in molecular testing using mixed-methods.

Using rigorous approaches proven successful in our prior work, we will recruit patient and clinician participants from each site to complete semi-structured interviews and structured questionnaires. The goal of this objective is to understand contextual mechanisms (e.g., patient, clinician, clinic, structural factors) shaping adoption, reach, and effectiveness of each intervention and identify how response may differ by key characteristics. These data will be analyzed using convergent mixed methods analysis, which employs the simultaneous collection and analysis of both quantitative and qualitative data to gain a comprehensive understanding of the multi-level factors shaping trial outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Participants with a histological, or cytological diagnosis of metastatic non-squamous (mNSq) non-small cell lung cancer (NSCLC) who have not yet received systemic treatment for metastatic disease.
* Participants must be seen at Lancaster General Health (LGH), Penn Presbyterian Medical Center (PPMC), Penn Medicine Cherry Hill (PMCH), Penn Medicine Princeton Health (PMPH), Penn Medicine Voorhees (PMV) or Penn Medicine Washington Township (PMWT) for mNSq NSCLC.

Exclusion Criteria:

* Participants with incomplete staging information.
* Children, pregnant women, fetuses, neonates, or prisoners are not included in this research study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2023-06-15 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Availability of comprehensive molecular test results prior to first line therapy for patients with newly diagnosed mNSq NSCLC | Measured up to 6 weeks from initial diagnosis
  Were comprehensive molecular test results available prior to initiation of 1L therapy? (Yes/No)

SECONDARY OUTCOMES:
Successful EHR based nudge delivery | Measured up to 6 weeks from randomization
  Amongst eligible patients, calculate the proportion of patients for whom the EHR nudge fired successfully (Yes/No). Applicable for the patients enrolled in the time periods following randomization.
Turnaround time of delivery of provider focused alerts | Measured up to 6 weeks from randomization
  Reported as number of days, median. Applicable for the patients enrolled in the time periods following randomization.
Completion of comprehensive molecular testing & modality used | Measured up to 3 months from initial diagnosis
  Relative and absolute change in completion of comprehensive testing by tissue and plasma, plasma alone, or tissue alone will be tabulated.
Reasons for failure to complete comprehensive molecular testing: | Measured up to 3 months from initial diagnosis
  Summarize reasons for failure of completion of testing i. Tissue related (QNS) ii. Patient related factors (unable to biopsy, patient declined biopsy etc.) iii. Assay related factors (plasma assay does not detect mutations) iv. Other
Time to molecularly informed treatment initiation | Measured up to 6 weeks from initial diagnosis
  i. Calculated as time to therapy from the date of diagnosis of Stage IV disease (date of biopsy) ii. Calculated as time to therapy from the date of first new patient visit with medical oncology
Type of therapy received | Measured up to 3 months from initial diagnosis
  i. Targeted therapy ii. Chemo-immunotherapy iii. Immunotherapy iv. Clinical trial or n v. None
Overall survival | Measured up to 1 year from the time of randomization to death from any cause
  i. Time from initial diagnosis to date of death or last follow up. ii. 1 year and 2-year overall survival rates will be calculated for the intervention group, and compared to baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Charu Aggarwal, MD, MPH, Principal Investigator — Penn Medicine
Locations (6):
- United States (6):
  - Penn Medicine Cherry Hill, Cherry Hill, New Jersey
  - Penn Medicine Princeton Health, Plainsboro, New Jersey
  - Penn Medicine Washington Township, Sewell, New Jersey
  - Penn Medicine Voorhees, Voorhees Township, New Jersey
  - Penn Medicine Lancaster General Health, Lancaster, Pennsylvania
  - Penn Presbyterian Medical Center, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No
A Clinical Study Report will be made available to the study sponsor.

REFERENCES:
- [Background] Aggarwal C, Rolfo CD, Oxnard GR, Gray JE, Sholl LM, Gandara DR. Strategies for the successful implementation of plasma-based NSCLC genotyping in clinical practice. Nat Rev Clin Oncol. 2021 Jan;18(1):56-62. doi: 10.1038/s41571-020-0423-x. Epub 2020 Sep 11. PMID 32918064
- [Background] Rolfo C, Mack P, Scagliotti GV, Aggarwal C, Arcila ME, Barlesi F, Bivona T, Diehn M, Dive C, Dziadziuszko R, Leighl N, Malapelle U, Mok T, Peled N, Raez LE, Sequist L, Sholl L, Swanton C, Abbosh C, Tan D, Wakelee H, Wistuba I, Bunn R, Freeman-Daily J, Wynes M, Belani C, Mitsudomi T, Gandara D. Liquid Biopsy for Advanced NSCLC: A Consensus Statement From the International Association for the Study of Lung Cancer. J Thorac Oncol. 2021 Oct;16(10):1647-1662. doi: 10.1016/j.jtho.2021.06.017. Epub 2021 Jul 8. PMID 34246791
- [Background] Singal G, Miller PG, Agarwala V, Li G, Kaushik G, Backenroth D, Gossai A, Frampton GM, Torres AZ, Lehnert EM, Bourque D, O'Connell C, Bowser B, Caron T, Baydur E, Seidl-Rathkopf K, Ivanov I, Alpha-Cobb G, Guria A, He J, Frank S, Nunnally AC, Bailey M, Jaskiw A, Feuchtbaum D, Nussbaum N, Abernethy AP, Miller VA. Association of Patient Characteristics and Tumor Genomics With Clinical Outcomes Among Patients With Non-Small Cell Lung Cancer Using a Clinicogenomic Database. JAMA. 2019 Apr 9;321(14):1391-1399. doi: 10.1001/jama.2019.3241. PMID 30964529
- [Background] Robert NJ, Espirito JL, Chen L, Nwokeji E, Karhade M, Evangelist M, Spira A, Neubauer M, Bullock S, Walberg J, Cheng SK, Coleman RL. Biomarker testing and tissue journey among patients with metastatic non-small cell lung cancer receiving first-line therapy in The US Oncology Network. Lung Cancer. 2022 Apr;166:197-204. doi: 10.1016/j.lungcan.2022.03.004. Epub 2022 Mar 10. PMID 35313244
- [Background] Thompson JC, Yee SS, Troxel AB, Savitch SL, Fan R, Balli D, Lieberman DB, Morrissette JD, Evans TL, Bauml J, Aggarwal C, Kosteva JA, Alley E, Ciunci C, Cohen RB, Bagley S, Stonehouse-Lee S, Sherry VE, Gilbert E, Langer C, Vachani A, Carpenter EL. Detection of Therapeutically Targetable Driver and Resistance Mutations in Lung Cancer Patients by Next-Generation Sequencing of Cell-Free Circulating Tumor DNA. Clin Cancer Res. 2016 Dec 1;22(23):5772-5782. doi: 10.1158/1078-0432.CCR-16-1231. Epub 2016 Sep 6. PMID 27601595
- [Background] Leighl NB, Page RD, Raymond VM, Daniel DB, Divers SG, Reckamp KL, Villalona-Calero MA, Dix D, Odegaard JI, Lanman RB, Papadimitrakopoulou VA. Clinical Utility of Comprehensive Cell-free DNA Analysis to Identify Genomic Biomarkers in Patients with Newly Diagnosed Metastatic Non-small Cell Lung Cancer. Clin Cancer Res. 2019 Aug 1;25(15):4691-4700. doi: 10.1158/1078-0432.CCR-19-0624. Epub 2019 Apr 15. PMID 30988079
- [Background] Aggarwal C, Thompson JC, Black TA, Katz SI, Fan R, Yee SS, Chien AL, Evans TL, Bauml JM, Alley EW, Ciunci CA, Berman AT, Cohen RB, Lieberman DB, Majmundar KS, Savitch SL, Morrissette JJD, Hwang WT, Elenitoba-Johnson KSJ, Langer CJ, Carpenter EL. Clinical Implications of Plasma-Based Genotyping With the Delivery of Personalized Therapy in Metastatic Non-Small Cell Lung Cancer. JAMA Oncol. 2019 Feb 1;5(2):173-180. doi: 10.1001/jamaoncol.2018.4305. PMID 30325992
- [Background] Shelton RC, Chambers DA, Glasgow RE. An Extension of RE-AIM to Enhance Sustainability: Addressing Dynamic Context and Promoting Health Equity Over Time. Front Public Health. 2020 May 12;8:134. doi: 10.3389/fpubh.2020.00134. eCollection 2020. PMID 32478025
- [Background] Rendle KA, Abramson CM, Garrett SB, Halley MC, Dohan D. Beyond exploratory: a tailored framework for designing and assessing qualitative health research. BMJ Open. 2019 Aug 27;9(8):e030123. doi: 10.1136/bmjopen-2019-030123. PMID 31462482
- [Background] Kane H, Lewis MA, Williams PA, Kahwati LC. Using qualitative comparative analysis to understand and quantify translation and implementation. Transl Behav Med. 2014 Jun;4(2):201-8. doi: 10.1007/s13142-014-0251-6. PMID 24904704
- [Background] Whitaker RG, Sperber N, Baumgartner M, Thiem A, Cragun D, Damschroder L, Miech EJ, Slade A, Birken S. Coincidence analysis: a new method for causal inference in implementation science. Implement Sci. 2020 Dec 11;15(1):108. doi: 10.1186/s13012-020-01070-3. PMID 33308250

DOCUMENTS (3):
  • Study Protocol: Revised iNUDGE Protocol 04.08.2025 (2025-04-08): https://cdn.clinicaltrials.gov/large-docs/87/NCT05853887/Prot_001.pdf
  • Study Protocol and Statistical Analysis Plan: Original Protocol 03.24.2023 (2023-03-24): https://cdn.clinicaltrials.gov/large-docs/87/NCT05853887/Prot_SAP_000.pdf
  • Statistical Analysis Plan: iNUDGE Statistical Analysis Plan 04.30.2025 (2025-04-30): https://cdn.clinicaltrials.gov/large-docs/87/NCT05853887/SAP_002.pdf